CLINICAL TRIAL: NCT00652730
Title: Comparative, Randomized, 3-Way Crossover Bioavailability Study of Par and Bristol-Myers Squibb (Buspar)15 mg Buspirone HCl Tablets Following Administration of a 30 mg Dose in Healthy Adult Males Under Fed and Fasting Conditions
Brief Title: Bioavailability Study of (Buspar) Buspirone HCl Tablets Under Fasting and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Phoenix International Life Sciences, Inc. (Industry)
Responsible Party: Alfred Elvin/Director of Biopharmaceutics, Par Pharmaceutical, Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 980564
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: To Determine Bioequivalence Under Fed Conditions
Keywords: bioequivalence; buspirone HCl; fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Buspirone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Subjects received the Par formulated product under fasting conditions
  Interventions: Drug: Buspirone HCl
- B (Experimental): Subjects received the Par formulated product under fed conditions
  Interventions: Drug: Buspirone HCl
- C (Active Comparator): Subjects received the Bristol-Myers Squibb formulated product under fed conditions
  Interventions: Drug: Buspar

INTERVENTIONS:
Drug: Buspirone HCl — Tablets, 30 mg, single-dose, fasting conditions
  Other Names: Buspar
  Arms: A
Drug: Buspirone HCl — Tablets, 30 mg, single-dose, fed conditions
  Other Names: Buspar
  Arms: B
Drug: Buspar — Tablets, 30 mg, single-dose, fed conditions
  Other Names: Buspirone HCl
  Arms: C

SUMMARY:
To compare the single-dose bioavailability of Par and Bristol-Myers Squibb Buspirone HCl Tablets

DETAILED DESCRIPTION:
To compare the single-dose bioavailability of Par and Bristol-Myers Squibb (Buspar) 15 mg buspirone HCl tablets, following administration of a 30 mg dose, under fed conditions. In addition, the bioavailability of the Par product was compared under fed and fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, 18-45 years of age
* Weighing at least 60 kg, who are within 10% of their ideal weights (Table of "Desirable Weights of Adults", metropolitan Life Insurance Company, 1983)
* Physical examination and laboratory tests of hematologic, hepatic and renal functions.
* Medically healthy subjects with clinically normal laboratory profiles will be enrolled in the study

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.
* In addition, the presence of alcoholism or drug abuse within the past year: hypersensitivity or idiosyncratic reaction to buspirone HCl.
* Subjects who have been receiving monoamine oxidase inhibitors.
* Subjects who have been on an abnormal diet (for whatever reason) during the 28 days preceding the study.
* Subjects who, through completion of the study, would have donated in excess of 500 mL blood in 14 days, or 500-750 mL blood in 14 days (unless approved by the Principal Investigator, 1000 mL blood in 90 days, 1250 mL blood in 120 days, 1500 mL blood in 180 days, 2000 mL blood in 270 days, 2500 mL blood in 1 year.
* Subjects who have participated in another clinical trial with 28 days of study start.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 1998-07; Primary Completion 1998-09 (Actual); Study Completion 1998-09 (Actual)

PRIMARY OUTCOMES:
Rate and extent of absorption | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Surfaty, MD, Principal Investigator — Phoenix International Life Sciences, Inc.
Locations (1):
- Phoenix International Life Sciences inc, Saint-Laurent, Quebec, Canada